CLINICAL TRIAL: NCT02116491
Title: Test of a Novel Visual Sputum Suctioning System in Mechanically Ventilated Patients
Brief Title: Visual Sputum Suctioning System Tests in Mechanically Ventilated Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Jinxing Wu, PhD, Professor, First Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JWu
Record Dates: First submitted 2014-04-12; First posted 2014-04-17 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Ineffective Airway Clearance; Respiratory Tract Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Closed suction system (No Intervention): All ES procedures were performed on indication by RICU nurses and according to protocol, according to which Cloesd suction system was performed which the patient remained connected to the ventilator. The catheter was inserted into the endotracheal tube until resistance was met and withdrawn 0.5 cm. A negative pressure of maximum 150mmHg was set, and the catheter was withdrawn while gently rotating. The procedure lasted for a total of 10 seconds. Nonsterile gloves were to be used during all procedures.
- Visual Sputum Suctioning System (Experimental): All ES procedures were performed on indication by RICU nurses and according to protocol, according to which Closed suction system was performed which the patient remained connected to the ventilator. The double-lumen catheter of the Visual Sputum Suctioning System integrated with a 0.9-mm micro-imaging fiber was inserted into the endotracheal tube until resistance was met and withdrawn 0.5 cm. A negative pressure of maximum 150mmHg was set, and the catheter was withdrawn while gently rotating. The procedure lasted for a total of 10 seconds. Nonsterile gloves were to be used during all procedures.
  Interventions: Device: Visual Sputum Suctioning System

INTERVENTIONS:
Device: Visual Sputum Suctioning System — All ES procedures were performed on indication by RICU nurses and according to protocol, according to which Closed suction system was performed which the patient remained connected to the ventilator. The double-lumen catheter of the Visual Sputum Suctioning System integrated with a 0.9-mm micro-imaging fiber was inserted into the endotracheal tube until resistance was met and withdrawn 0.5 cm. A negative pressure of maximum 150mmHg was set, and the catheter was withdrawn while gently rotating. The procedure lasted for a total of 10 seconds. Nonsterile gloves were to be used during all procedures.
  Other Names: VSSS
  Arms: Visual Sputum Suctioning System

SUMMARY:
BACKGROUND: The investigators developed a fiber-optic-guided endotracheal suction catheter (visual sputum suctioning system or VSSS), which the investigators previously tested in vitro and animals. It integrates a 0.9-mm micro-imaging fiber into a 3.7-mm double-lumen catheter.

PURPOSE: The purpose of this study was to investigate the safety and efficacy of sputum suctioning system in mechanical ventilated patients in respiratory intensive care unit (RICU). The investigators compare the weight of secretions collected, vital signs, and tracheal wall injury between two groups of patients randomized to have VSSS combined with closed system suction (CSC) suction and patients having CSC suction alone.

HYPOTHESIS: The investigators theorized that the VSSS collected more sputum and caused less change of vital signs than conventional CSC.

DETAILED DESCRIPTION:
Study design: This is a randomized controlled trial study, including patients ventilated in one respiratory intensive care unit (RICU). Two suction systems (The novel VSSS and conventional CSS alone) will be compared at time point before (baseline), immediately after, 3 min after, and 5 min after suctioning.

Background: Sputum suctioning is a routine clinical procedure that is crucial for keeping the airway open, to reduce the incidence of respiratory-tract infections. In most circumstances, a conventional catheter with a single-lumen channel is used for sputum suctioning. However, this procedure Involves blind manipulation of the catheter on the part of the clinician and thus depends largely on the clinician's skills and experience. Therefore, complications occur in some patients, especially on the changes of the parameters of the heart-lung system. In addition, because clinicians cannot directly target sputum in the trachea, the efficiency of the procedure may be reduced.

Recently, a visual sputum suctioning system (VSSS) was developed in our research group. It integrates a 0.9-mm micro-imaging fiber into a 3.7-mm double-lumen catheter.

In vitro tests investigators found that the ability to visualize the airway allows targeting of sputum, which compensates for the smaller lumen and makes the suctioning procedure more efficient overall. In addition, in animal tests investigators found that the VSSS collected more sputum and caused less tracheal mucosa damage than conventional suctioning.

Purpose: The present study investigated the safety and efficacy of sputum suctioning system with this double-lumen catheter in mechanical ventilated patients in respiratory intensive care unit (RICU). The purpose of this study was to compare the weight of secretions collected, vital signs, and tracheal wall injury between two groups of patients randomized to have VSSS combined with closed system suction (CSC) suction and patients having CSC suction alone. investigators theorized that the VSSS collected more sputum and caused less change of vital signs than conventional CSC.

Registry procedure: All requested information will be recorded on case report forms and explanation will be reported for any missing data. False data will be clearly corrected, and signed by investigator or authorized person.

Monitoring will be realized by the co-investigator in association with the clinical research associate.

Sample size assessment: Number of subjects: 40 patients. Three months should be necessary to include these patients.

Statistical analysis: Investigators determined that 20 patients per group would provide a power of 95%, with a α level of 5%.

Results will be expressed as means ± Standard Deviation. SPSS 10.0 (Chicago, Illinois, USA) for the statistical calculation was used. P values < 0.05 were considered statistically significant. Investigators used the nonparametric t test for normally distributed data, and the nonparametric Wilcoxon-Mann-Whitney rank test for other data.Investigators used repeated-measures analysis of variance at four time points (before suctioning, immediately after suctioning, 3 min after suctioning, and 5 min after suctioning) to analyze changes and differences in PaO2, heart rate, and mean arterial pressure.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to RICU
* 18 years old or more
* Ventilated more than 24 hours mechanical ventilation
* Patients with stability (MAP>70 mmHg, HR<130 b/min)
* Signed informed consent

Exclusion Criteria:

* Current or past participation in another intervention trial conflicting with the present study patients with stupor and coma
* Any clinical events or practitioner interventions within 15 min prior to study enrollment (eg, a change in ventilator settings, hemodynamic instability [DBP >100 mmHg; ↑or 20mmHg in PaO2; ↑20 b/min in HR]; sever hypoxemia [SpO2<85%, PaO2<50mmHg])
* Had heart or lung or heart transplantation.
* Had massive hemoptysis.
* Pregnant women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-05 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in hemodynamic and respiratory data at 5 min | Patients will be followed until 2 hour after suction.
  The hemodynamic and respiratory data including heart rate, arterial partial pressure of oxygen and mean arterial pressure will be recorded before (baseline), immediately after, 3 min after, and 5 min after suctioning.
Rate of hemorrhage | Patients will be followed until 2 hour after suction.

SECONDARY OUTCOMES:
Weight gain of the suction catheter | Until finished suctioning (An expected average of 10 min)
  Weight gain of the suction catheter due to secretions will be measured by mean of a high precision laboratory scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jinxing Wu, PhD, Pro, Study Chair — Department of Respiratory Medicine, First Affiliated Hospital of Chongqing Medical University, Chongqing, China
Locations (1):
- Department of Gerontology, First Affiliated Hospital of Chongqing Medical University,, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Background] Choi JS, Jones AY. Effects of manual hyperinflation and suctioning in respiratory mechanics in mechanically ventilated patients with ventilator-associated pneumonia. Aust J Physiother. 2005;51(1):25-30. doi: 10.1016/s0004-9514(05)70050-7. PMID 15748122
- [Background] Yorioka K, Oie S, Kamiya A. Microbial contamination of suction tubes attached to suction instruments and preventive methods. Jpn J Infect Dis. 2010 Mar;63(2):124-7. PMID 20332576
- [Background] Barnes CA, Kirchhoff KT. Minimizing hypoxemia due to endotracheal suctioning: a review of the literature. Heart Lung. 1986 Mar;15(2):164-76. No abstract available. PMID 3512492
- [Background] Brochard L, Mion G, Isabey D, Bertrand C, Messadi AA, Mancebo J, Boussignac G, Vasile N, Lemaire F, Harf A. Constant-flow insufflation prevents arterial oxygen desaturation during endotracheal suctioning. Am Rev Respir Dis. 1991 Aug;144(2):395-400. doi: 10.1164/ajrccm/144.2.395. PMID 1859066
- [Background] Maggiore SM, Lellouche F, Pigeot J, Taille S, Deye N, Durrmeyer X, Richard JC, Mancebo J, Lemaire F, Brochard L. Prevention of endotracheal suctioning-induced alveolar derecruitment in acute lung injury. Am J Respir Crit Care Med. 2003 May 1;167(9):1215-24. doi: 10.1164/rccm.200203-195OC. Epub 2003 Feb 13. PMID 12615633
- [Background] Almgren B, Wickerts CJ, Heinonen E, Hogman M. Side effects of endotracheal suction in pressure- and volume-controlled ventilation. Chest. 2004 Mar;125(3):1077-80. doi: 10.1378/chest.125.3.1077. PMID 15006972